CLINICAL TRIAL: NCT05021276
Title: A Prospective Multicenter, Single-arm Clinical Study of Anti-CD25 Monoclonal Antibody Combined With Ruxolitinib in the Treatment of Grade 3-4 Steroid-resistant Acute Graft-versus-host Disease
Brief Title: Basiliximab Combined With Ruxolitinib as Second-line Treatment of Grade 3-4 Steroid-resistant aGVHD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Soochow Hopes Hematonosis Hospital (Unknown); The Second People's Hospital of Huai'an (Other)
Responsible Party: Principal Investigator, Xuefeng He, chief physician, The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GVHD-001
Record Dates: First submitted 2021-08-17; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Safety and Efficacy
MeSH Terms: interventions — ruxolitinib; Basiliximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ruxolitinib+basiliximab (Experimental): Patients with grade 3-4 steroid-refractory aGVHD receive combined therapy of basiliximab and ruxolitinib.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib and basiliximab are both second-line treatment for grade 3-4 steroid-resistant acute graft-versus-host disease.
  Other Names: basiliximab

SUMMARY:
Acute graft-versus-host disease (aGVHD) is the most common life-threatening complication of allogeneic hematopoietic stem cell transplantation. The recognized first-line treatment for grade 3-4 aGVHD is systemic glucocorticoid. However, there is no recognized second-line treatment for grade 3-4 steroid-resistant aGVHD (SR-aGVHD). The investigators try to observe the efficacy and safety of early application of anti-CD25 monoclonal antibody(basiliximab) combined with ruxotilinib in the treatment of severe SR-aGVHD.

DETAILED DESCRIPTION:
Adults ages 18-65 with grade 3-4 SR-aGVHD

Design

Participants with grade 3-4 steroid-refractory acute GVHD (progression after 3 days or lack of improvement after 5 days of 1.5-2 mg/kg/d systemic steroids) receive combined therapy of basiliximab and ruxolitinib.

Basiliximab is given 20mg twice a week for week 1, and then once a week until GVHD of the participants reaches grade 1(3 episodes for minimum).

Ruxolitinib is given 5mg twice a day for one day and then escalates to 10mg twice a day if the participant is not administered with triazole antifungal agent.

The drug dose will be adjusted according to participants' clinical manifestations, blood cell count, infection status and so on.

For participants with lower gastrointestinal GVHD, intravenous cyclosporine or tacrolimus is given and plasma concentration is monitored in a safe and effective range.

Best supportive treatment is given, including broad-spectrum anti-infection, nutrition support, and blood transfusion.

The investigators access the efficacy and safety of second-line therapy once a week from day 14 until complete remission is received. Then the investigators access the hematological disease status, aGVHD, cGVHD, infection state once a month.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary grade 3-4(according to MAGIC criteria) steroid-resistant acute graft-versus-host disease(progression after 3 days or lack of improvement after 5 days of systemic 1.5-2 mg/kg steroids).
* Age 18-65.
* ECOG score≤3.
* Must be able to understand and willing to participate in the study and sign the informed consent.

Exclusion Criteria:

* Refractory/secondary graft-versus-host disease.
* Severe complications such as myocardial infarction, chronic cardiac insufficiency, hepatic failure, renal insufficiency, etc.
* Clinically uncontrolled active infections.
* Other Malignant tumors with progression.
* Ecg: QT interval > 450 ms.
* Allergic to arsenic agent.
* Pregnant or lactating women.
* Expected survival <60 days.
* Undergoing other drug clinical trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
overall response rate at day 28 | day 28
  The primary endpoint is the overall response rate (ORR) at day 28 defined as proportion of patients demonstrating partial (PR) or complete response (CR) without requirement for additional systemic immunosuppressive therapy (IST) at day 28 after second-line treatment initiates.

SECONDARY OUTCOMES:
ORR at d14/d56 | day 14, day 56
  overall response rate at day 14/56
Time to response | through study completion(median 12 days according to previous study)
  Time to response, defined as time from the day treatment initiates to the date of first documentation PR or CR.
Duration of response | through study completion, an average of 1year
  Duration of response, assessed for responders only by calculating the time from first response to the date of first observation of aGvHD relapse/progression or the date of additional IST for GvHD.
OS | through study completion, an average of 1year
  Overall survival (OS) defined as time from the day treatment initiates to the date of death from any cause.
EFS | through study completion, an average of 1year
  Event-free survival (EFS) defined as the time from the day treatment initiates to the date of recurrence of underlying hematologic disease, graft failure or death due to any cause.
incidence rate of secondary grade 3-4 liver aGVHD | through study completion, an average of 1 year
  incidence rate of secondary grade 3-4 liver aGVHD
incidence rated of chronic GVHD | through study completion, an average of 1 year
  incidence rated of chronic GVHD

CONTACTS AND LOCATIONS:
Overall Officials: Xuefeng He, doctor, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou F, Pan T, Li X, Du F, Ma X, Zhang Y, Wu D, Han Y, Xue S, Miao M, Tao T, He X, Chen S. Exploration of efficacy and safety of combined therapy of basiliximab with ruxolitinib for grade 3-4 steroid-refractory acute graft-versus-host disease: a registered clinical trial (NCT05021276). Bone Marrow Transplant. 2023 Aug;58(8):959-961. doi: 10.1038/s41409-023-02005-4. Epub 2023 May 30. No abstract available. PMID 37253803